CLINICAL TRIAL: NCT05393609
Title: Quality of Life and Surgery in Diverticular Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Life with diverticular disease
Record Dates: First submitted 2022-05-11; First posted 2022-05-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Diverticulitis Colon; Quality of Life; Diverticular Disease of Left Side of Colon
MeSH Terms: conditions — Diverticulitis, Colonic | interventions — Conservative Treatment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sigmoidectomy: Patients with diverticular disease undergoing elective resection of the sigmoid colon
  Interventions: Procedure: Sigmoidectomy
- Conservative: Patients with diverticular disease not referred to surgery, but conservative treatment
  Interventions: Dietary Supplement: Conservative

INTERVENTIONS:
Procedure: Sigmoidectomy — Conventional laparoscopic resection of the sigmoid colon
  Groups: Sigmoidectomy
Dietary Supplement: Conservative — According to current practice including advice on supplementary dietary fiber, analgetics, or laxatives when indicated.
  Groups: Conservative

SUMMARY:
Diverticular disease is one of the most common diseases of the gastrointestinal tract in industrial countries. Prevalence and admission rate due to diverticular disease increases.

Symptomatic patients usually present with acute uncomplicated or complicated diverticulitis. Recurrence rates of complicated diverticulitis are estimated to 10-30%. Recurrences, chronic complications or persisting pain, here collectively referred to as chronic diverticular disease, may be treated by elective sigmoidectomy. Currently, there is no specific criteria for elective surgery, but only a recommendation of a tailored approach depending on the patient's symptoms.

It is well established that diverticular disease has a negative impact on quality of life (QoL). Elective laparoscopic sigmoidectomy may increase QoL.

In this prospective study, we will prospectively examine QoL, patient-related outcomes and peri- and postoperative outcome of elective sigmoidectomy for chronic diverticular disease, and compare it to conservatively treated patients.

DETAILED DESCRIPTION:
Design: Prospective, multicentre, observational

Locations: Hospitals in Central and Northern Denmark Region (6 hospitals).

Time: Recruitment starts in April 2022 and is planned to be completed in 2024.

Patients: All patients referred to a surgical clinic due to chronic diverticular disease.

Allocation for surgery or conservative treatment: Patients will be treated according to Danish National Guidelines for treatment of diverticular disease. The study will not influence the treatment of the patient, but only observe and evaluate current daily practice.

Intervention: Patients will be asked to answer questionnaires at inclusion and again after 1 year. Patients treated with sigmoidectomy will also be asked to answers questionnaires 3 weeks and 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Referred to surgical clinic due to diverticular disease
* Colonic diverticula verified by CT or endoscopy

Exclusion Criteria:

* Previous colonic resection other than appendectomy
* Previous or current colorectal cancer
* Previous or current disseminated cancer
* Inflammatory bowel disease
* Psychiatric disorder influencing the ability to answer questionnaires
* Inadequate Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with recurrent or chronic diverticular disease referred to a surgical department in Central or Northern Denmark Region.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Change from baseline to 1 year follow-up.
  Gastrointestinal Quality of Life (GIQLI) 36 items. Total score 0-144 (0=worst, 144=best).
Disease-specific quality of life | Baseline.
  Diverticulitis quality of life (DV-QoL) 16 items. Total score 0-10 (0= best,10=worst).

SECONDARY OUTCOMES:
Generic quality of life | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  EuroQol-5 Domain 5-level (EQ-5D-5L) 5 items. Total score 5-25 (5=best. 25 = worst). Visual analog scale 0-100 (0=worst, 100= best).
Bowel function | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  Patient-assessment of constipation symptoms (PAC-SYM) 12 items. Total score 0-50 (0=best, 50=worst).
Bowel function | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  Low anterior resection syndrome score (LARS score) 5 items. Total score 0-42 (0=best, 42=worst).
Pain related to diverticular disease | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  Modified Rectal Cancer Pain Score 7 items. Total score 0-45 (0= best, 45= worst). 7 item. Total score 0-29 (0= worst, 65= best).
Urinary dysfunction - females | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  International Consultation on Incontinence Questionnaire Female Lower Urinary Tract Symptoms (CIQ-FLUTS) 13 items. Total score 0-52 (0=best, 52=worst).
Urinary dysfunction - males | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  International Consultation on Incontinence Questionnaire Male Lower Urinary Tract Symptoms (ICIQ-MLUTS) 14 items. Total score 0-56 (0=best, 56=worst).
Sexual dysfunction - females | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  Modified Rectal Cancer Female Sexuality Score 7 items. Total score 0-29 (0=best, 29= worst). 14 item. Total score 0-56 (0=best, 56=worst).
Sexual dysfunction - males | Change from baseline to 3 weeks follow-up, 3 months follow-up and 1 year follow-up.
  The International Index of Erectile Function Questionnaire (IIEF) 15 items. Total score 0-65 (0= worst, 65= best).
Postoperative morbidity | 30 days
  Postoperative complications classified according to the Clavien-Dindo classification
Postoperative mortality | 30 days
  Mortality within the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Helene R Dalby, MD, Principal Investigator — Randers Regional Hospital
Locations (1):
- Randers Regional Hospital, Randers, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No